CLINICAL TRIAL: NCT04304495
Title: GAPcare II: The Geriatric Acute & Post-acute Care Coordination Program for Fall Prevention in the Emergency Department
Brief Title: The Geriatric Acute & Post-acute Care Coordination Program for Fall Prevention in the Emergency Department II
Acronym: GAPcareII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Apple Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 22-2089; K76AG059983 (NIH)
Record Dates: First submitted 2019-12-06; First posted 2020-03-11 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Fall
Keywords: prevention; emergency department; digital health; Apple Watch; physical therapy; pharmacy; GAPcare; Geriatric
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants will be randomly assigned (by the REDCap program) 1:1 to the intervention or usual care arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): In addition to the usual care arm, the Intervention arm will receive a physical therapy and pharmacy consultation in the ED. PTs will perform a fall risk assessment and provide recommendations on the safety of discharge. Pharmacists will perform medication review, recommend cessation or tapering of medication that increase fall risk using motivational interviewing (MTM) techniques.
  The participants will also receive Apple Watch training and an Apple Watch to perform tasks that test their memory and mobility during their ED visit and during our home visits at 1,3, 6, and 12 month after enrollment.
  Interventions: Other: Fall Prevention
- Usual care arm (No Intervention): The ED clinician will perform a standard medical evaluation, including a focused history and exam to identify injuries, laboratory tests and radiologic imaging. If necessary, the patient will receive consultation with specialty services (e.g., orthopedics).
  The participants will also receive Apple Watch training and an Apple Watch to perform tasks that test their memory and mobility during their ED visit and during our home visits at 1,3, 6, and 12 month after enrollment.

INTERVENTIONS:
Other: Fall Prevention — The intervention arm participants will receive a physical therapy and pharmacy consults as well as Apple Watch training and an Apple Watch device to test memory and mobility during the ED visit and during our home visits.
  Arms: Intervention

SUMMARY:
In brief, this K76 study consists of a small open trial to refine the study protocol and train study personnel on study procedures (Aim 1.b.). In Aim 2, we will recruit older adults into a multidisciplinary fall prevention pilot study. Participants will be randomly assigned to usual care with a traditional fall evaluation by an ED clinician (i.e., ED medical staff member) or an intervention. In the intervention, participants will receive an in-ED consultation by a physical therapist and pharmacist to determine reasons for the fall and offer additional education and training. Participants will be provided an Apple Watch to record measures of fitness and falls, if possible, in the following 12 months. Recurrent falls will be measured in twelve-month follow-up.

DETAILED DESCRIPTION:
In order to determine whether a multifactorial fall prevention intervention is feasible, acceptable and may reduce recurrent falls in older adults presenting to the ED after a fall, we will randomize patients to usual care with a traditional fall evaluation by an ED clinician or an intervention. Patients in the intervention arm receive a fall risk assessment and recommendations by a physical therapist. They are also evaluated by a pharmacist and participate in a medication therapy management session with the aim to reduce fall risk increasing medication.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling adult (non-institutionalized) 65 years-old or older presenting to ED after a fall
* Fall not due to syncope or external force (i.e., struck by car or assault)
* Fall not due to serious illness (i.e., stroke, acute myocardial infarction)
* Will be discharged to home/assisted living/rehabilitation at completion of ED visit (i.e., not admitted)
* Legally authorized representative able to give informed consent if patient has cognitive impairment on Six Item Screener (score of less than four) either over the phone with witness present or in person
* Must screen or test negative for COVID-19

Exclusion Criteria:

* Unable to give informed consent due to intoxication or altered mental status
* Presence of injuries that prevent mobilization (i.e., pelvic or lower extremity fractures)
* Allergies to any wearable device component
* Unable or unwilling to wear Apple Watch at home (only for periodic study visits)
* Patient has advanced cancer and/or is on hospice care
* Pts coming from SNF or nursing home
* Previously enrolled in GAPcare II Aim1.b

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 197 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2025-02-02 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
Rate of study activity completion | 12 months
  Rate of participants who completed all study activities, including initial enrollment and multiple follow up visits over a 12 month period

SECONDARY OUTCOMES:
Change in gait speed | 12 months
  Apple watch determined; average change in gait speed over 12-month follow-up
Change in activity level | 12 months
  Apple watch determined; average change in proportion of time spent active per day (e.g. walking, running, not driving or sedentary)
Number of recurrent falls | 12 months
  Number of falls in person months
Number of ED re-visits | 12 months
  Any visit to the ED in the 12-month follow-up
Rate of hospitalization | 12 months
  Any hospital admission in the 12-month follow-up
Rate of permanent moves to nursing homes | 12 months
  Any move to a nursing home for >30 days
Mortality rate | 12 months
  All cause patient mortality in follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M Goldberg, MD, ScM, Principal Investigator — University of Colorado, Denver
Locations (3):
- United States (3):
  - University of Colorado Hospital, Aurora, Colorado
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island

REFERENCES:
- [Background] Strauss DH, Davoodi NM, Healy M, Metts CL, Merchant RC, Banskota S, Goldberg EM. The Geriatric Acute and Post-Acute Fall Prevention Intervention (GAPcare) II to Assess the Use of the Apple Watch in Older Emergency Department Patients With Falls: Protocol for a Mixed Methods Study. JMIR Res Protoc. 2021 Apr 1;10(4):e24455. doi: 10.2196/24455. PMID 33792553